CLINICAL TRIAL: NCT06053307
Title: Treating Psychosocial Distress in Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00108155; R00EY033027 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma, Primary Open Angle; Distress, Emotional; Anxiety; Depression
MeSH Terms: conditions — Glaucoma, Open-Angle; Anxiety Disorders; Depression | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VISION-ACT: Acceptance commitment therapy via a mobile-application (Experimental): The arm will pilot a behavioral intervention to treat psychosocial distress in patients with glaucoma using acceptance commitment therapy (ACT) delivered via a mobile-application, called VISION-ACT. The intervention will be developed and refined using qualitative feedback from glaucoma patients and healthcare stakeholders.
  Interventions: Behavioral: Acceptance commitment therapy

INTERVENTIONS:
Behavioral: Acceptance commitment therapy — The baseline intervention will use ACT, a psychological intervention based on modern behavioral psychology, including relational frame theory, that uses acceptance and mindfulness strategies, along with commitment and behavior-change strategies to increase psychological flexibility. The proposed intervention will be delivered over a 6-week period, with each week including content related to one of the six tenets of ACT: cognitive defusion, acceptance, contact with the present moment, the observing self, values, and committed action. Each week will include educational material, skills work, and homework. The intervention will be delivered via a mobile application.

SUMMARY:
In this study, using three phases, the investigators will use an iterative development approach to refine a behavioral intervention for managing concomitant psychosocial distress in glaucoma. Phase 1: The investigators will begin by developing a baseline intervention using strategies from Acceptance and Commitment Therapy (ACT), and delivered using a mobile application. Phase 2: The investigators will refine the baseline intervention for glaucoma patients using qualitative interviews conducted with primary open-angle glaucoma (POAG) patients with psychosocial distress (N=20), and health professionals (N=5). Phase 3: Finally, the investigators will measure acceptability and feasibility of the refined intervention through a single-armed pilot study (N=25). The investigators hypothesize that the refined intervention will yield an acceptable and feasible intervention in a POAG patient population, setting the stage for a future efficacy study.

ELIGIBILITY:
Inclusion Criteria

* diagnosed with mild, moderate, or severe chronic glaucoma (e.g., POAG),
* had a visual field within the past year at the main Duke Eye Center,
* been prescribed pressure lowering eye drop medication,
* at least mild distress (based on PHQ-4),
* 18 years old,
* able to understand, speak, and read English, and
* be able to provide informed consent.

Exclusion Criteria

* diagnosed with borderline glaucoma or as a glaucoma suspect,
* had a glaucoma surgery in past month (e.g., trabeculectomy, glaucoma drainage device/tube),
* visual acuity of worse than 20/70 in the better seeing eye,
* diagnosed with a major medical conditions (e.g., cancer, or another visual disorder, like macular degeneration),
* diagnosed with a psychiatric conditions (e.g., schizophrenia, bipolar disorder), and
* reported or suspected cognitive impairment indicated by provider or chart review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in psychosocial distress | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using the Hospital Anxiety and Depression Scale (HADS). The scale ranges from 0-42 with higher values indicating higher distress.
Change in psychosocial distress | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using the Subjective Unit of Distress (SUDS) scale. The scale ranges from 0-10 with higher values indicating higher distress.
Change in vision-related quality-of-life (QoL) | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using the National Eye Institute (NEI)- Visual Functioning Questionnaire (VFQ) 9. The scale ranges from 0-100 with higher values indicating higher vision-related QoL.
Change in health-related QoL | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using the CDC Health-Related Quality-of-Life 4-Item Scale. For our outcome we will use the self-rated scale from Poor to Excellent, which has a scale from 1-5, with higher values indicating higher QoL.

SECONDARY OUTCOMES:
Change in psychological flexibility | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using the Acceptance and Action Questionnaire 7-Item Scale. The scale ranges from 0-49 with higher values indicating lower psychological flexibility.
Change in disease acceptance | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using the Acceptance of Illness 8-Item Scale. The scale ranges from 8-40 with higher scores indicating better acceptance of illness.
Change in self-efficacy | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using Self-efficacy for managing chronic disease 6-Item Scale. The scale ranges from 6-60 with higher values indicating higher self-efficacy.
Change in mindfulness | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) 10-Item. The scale ranges from 10-40 with higher values indicating higher mindfulness.
Change in perceived social support | Measures will be administered at baseline (A1), immediately post-intervention (A2), and 1-month post treatment assessment (A3).
  Measured using 8-item Medical Outcomes Study Social Support Survey. The scale ranges from 8-40 with higher values indicating higher perceived social support.

OTHER OUTCOMES:
Study feasibility | Collected within a one-year period from the beginning of recruitment.
  Reaching target accrual (N=25) within a 12-month study recruitment period.
Study feasibility | Collected at the post-intervention assessment (A2), six-weeks after the initial assessment.
  <20% study attrition, defined as the percentage of participants who completed the post-intervention A2 assessment (primary end-point).
Study acceptability | Collected at the post-intervention assessment (A2), six-weeks after the initial assessment.
  ≥80% of participants reporting intervention satisfaction (i.e., Client Satisfaction Questionnaire mean≥3.00/4.00). The score ranges from 8 to 32, with larger numbers indicating greater satisfaction.
Study acceptability | Collected at the post-intervention assessment (A2), six-weeks after the initial assessment.
  ≥75% of participants reporting use of skills or ideas from the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Except for personal identifying data such as name, address and contact information, all raw survey and qualitative data, the data dictionary, and any statistical programs used to analyze the survey data will be preserved and shared. The rationale is to provide scientific collaborators with access to all data collected during the study while preserving participant privacy. The data will be shared through the NEI Data Commons.
Supporting Information: Study Protocol, Analytic Code